CLINICAL TRIAL: NCT02792972
Title: Antiseptic and Analgesic Action Acmella Oleracea Skin: Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ana Beatriz Alkimim Teixeira Loyola (Other)
Responsible Party: Sponsor-Investigator, Ana Beatriz Alkimim Teixeira Loyola, MD, Universidade do Vale do Sapucai
Organization: Universidade do Vale do Sapucai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Carol2014
Record Dates: First submitted 2016-05-23; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: Phythoterapy; Venipuncture Site Numbness; Antimicrobial; Analgesic
Keywords: Analgesic; Medicinal plants; Skin; Antimicrobial agents; Pain Measurement
MeSH Terms: interventions — Ethanol

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Acmella oleracea (Active Comparator): The plant extract A. oleracea manipulated with Transcutol® were used in the volunteers 3 minutes before the venipuncture
  Interventions: Other: A. oleracea
- alcohol 70% (Placebo Comparator): 70% alcohol were used in the volunteers 3 minutes before the venipuncture
  Interventions: Other: 70% alcohol

INTERVENTIONS:
Other: A. oleracea — The plant extract A. oleracea manipulated with Transcutol® were used in the volunteers before the venipuncture procedure as allocation in study groups. Held collection of skin microbiota by the swab technique and the end of the venipuncture procedure was applied to the volunteer, the visual numeric scale (VNS) standard to determine the degree of pain.
  Other Names: medical plants
  Arms: Acmella oleracea
Other: 70% alcohol — 70% alcohol were used in the volunteers before the venipuncture procedure as allocation in study groups. Held collection of skin microbiota by the swab technique and the end of the venipuncture procedure was applied to the volunteer, the visual numeric scale (VNS) standard to determine the degree of pain.
  Arms: alcohol 70%

SUMMARY:
Context: Research on natural products with therapeutic, analgesic or antimicrobial purpose should be encouraged to create new drugs. Acmella oleracea, typical plant of the Northern region of the country and popularly known as jambu, has aroused the interest of researchers because of its therapeutic potential. Objective: To evaluate the potential topical analgesic and antimicrobial of Acmella oleracea plant extract from the skin antisepsis in venipuncture procedures. Methods: This is a clinical, randomized, controlled trial with healthy volunteers recruited at the Clinic I of the collection of biological materials sector of the Hospital das Clinicas Samuel Libânio, in Pouso Alegre-MG. The plant extract A. oleracea manipulated with Transcutol® and 70% alcohol were used in the volunteers before the venipuncture procedure as allocation in study groups. Held collection of skin microbiota by the swab technique and the end of the venipuncture procedure was applied to the volunteer, the visual numeric scale (VNS) standard to determine the degree of pain.

DETAILED DESCRIPTION:
Context: Research on natural products with therapeutic, analgesic or antimicrobial purpose should be encouraged to create new drugs. Acmella oleracea, typical plant of the Northern region of the country and popularly known as jambu, has aroused the interest of researchers because of its therapeutic potential. Objective: To evaluate the potential topical analgesic and antimicrobial of Acmella oleracea plant extract from the skin antisepsis in venipuncture procedures. Methods: This is a clinical, randomized, controlled trial with healthy volunteers recruited at the Clinic I of the collection of biological materials sector of the Hospital das Clinicas Samuel Libânio, in Pouso Alegre-MG. The plant extract A. oleracea manipulated with Transcutol® and 70% alcohol were used in the volunteers before the venipuncture procedure as allocation in study groups. Held collection of skin microbiota by the swab technique and the end of the venipuncture procedure was applied to the volunteer, the visual numeric scale (VNS) standard to determine the degree of pain.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* without restriction as to ethnicity
* educational level and social class who agreed to participate by signing the Informed Consent and Informed (IC )

Exclusion Criteria:

* pregnant women (due to contractile properties that can cause )
* cancer patients
* chronic and refusal to participate in the study kidney

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The degree of pain in 15 healthy volunteers will be measured by the visual numeric scale (VNS) standard immediately after the venipuncture procedure. | 1 day
The skin microflora in 15 healthy volunteers will be measured counted the microorganism isolated by swab technique and plated on plates containing the medium Standard Methods Agar (PCA). | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Ana Beatriz A Teixeira Loyola, doctor, Study Director — Universidade do Vale do Sapucaí

IPD SHARING:
Plan to Share IPD: Undecided